CLINICAL TRIAL: NCT06160271
Title: Pilot Study of Liver Fibrosis Stage Assessment by Tep Fibroblast Activation Protein Imaging (68Ga-FAPI-46 TEP/TDM) in Patients With Biopsy for Suspected or Proven Nonalcoholic Steatohepatitis (NASH)
Brief Title: Study of Liver Fibrosis Stage Assessment by Fibroblast Activation Protein Imaging in Patients With Biopsy for Suspected or Proven Nonalcoholic Steatohepatitis
Acronym: HEFITEP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Elodie CHEVALIER, MD, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022PI044
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-11

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEP 68Ga-FAPI (Experimental): Use of a positron emission tomograph equipped with an X-ray scanner (PET/CT), essential for recording images after injection of a positron-emitting radiopharmaceutical (in this study, 68Ga-FAPI-46).
  Interventions: Drug: PET scan of 68Ga-FAPI

INTERVENTIONS:
Drug: PET scan of 68Ga-FAPI — Use of a positron emission tomograph equipped with an X-ray scanner (PET/CT), essential for recording images after injection of a positron-emitting radiopharmaceutical (in this study, 68Ga-FAPI-46).

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD), estimated to be 17% prevalent in France, can lead to non-alcoholic steatohepatitis (NASH), which in turn can progress to fibrosis, the ultimate stage of which is cirrhosis, a major cause of liver transplantation. The prevalence of NASH is increasing worldwide, along with that of type 2 diabetes and obesity. Significant liver fibrosis is estimated to affect at least 2.6% of the adult population in France.

The prognosis of patients with NASH is directly linked to the stage of liver fibrosis determined by biopsy, and these biopsies must now be repeated to assess the effect of treatments. Hepatic fibrosis is traditionally classified into five stages, from the absence of fibrosis (F0) to severe cirrhosis (F4), and passage from one stage to another is considered to demonstrate significant variation, likely to impact prognosis.

However, liver biopsy is painful. It can only analyze a very small proportion of liver volume (1/50,000), whereas the distribution of fibrosis is generally heterogeneous. Above all, biopsy is not devoid of risks, primarily hemorrhage, which can sometimes be severe or even fatal.

In line with current recommendations, clinical-biological algorithms, as well as ultrasound elastography or MRI, are used to assess the risk of fibrosis and the value of a liver biopsy. Generally speaking, these tests have the advantage of very good negative predictive values, making it possible to exclude the possibility of significant fibrosis in a large proportion of patients. However, their positive predictive values are weaker, even when these tests are combined. Above all, they do not allow us to follow the evolution of the fibrosis stage over time. This is why liver biopsies remain indispensable for determining the stage and severity of hepatic fibrosis and monitoring its evolution. It is therefore essential to develop more precise, non-invasive methods for accurately assessing the extent of liver fibrosis. This is the objective of the FreSH national cohort, which uses conventional biological techniques and in which our patients will also be included.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD), estimated to be 17% prevalent in France, can lead to non-alcoholic steatohepatitis (NASH), which in turn can progress to fibrosis, the ultimate stage of which is cirrhosis, a major cause of liver transplantation. The prevalence of NASH is increasing worldwide, along with that of type 2 diabetes and obesity. Significant liver fibrosis is estimated to affect at least 2.6% of the adult population in France The prognosis of patients with NASH is directly linked to the stage of liver fibrosis determined by biopsy, and these biopsies must now be repeated to assess the effect of treatments. Hepatic fibrosis is traditionally classified into five stages, from the absence of fibrosis (F0) to severe cirrhosis (F4), and passage from one stage to another is considered to demonstrate significant variation, likely to impact prognosis.

However, liver biopsy is painful. It can only analyze a very small proportion of liver volume (1/50,000), whereas the distribution of fibrosis is generally heterogeneous. Above all, biopsy is not devoid of risks, primarily hemorrhage, which can sometimes be severe or even fatal.

In line with current recommendations, clinical-biological algorithms, as well as ultrasound elastography or MRI, are used to assess the risk of fibrosis and the value of a liver biopsy. Generally speaking, these tests have the advantage of very good negative predictive values, making it possible to exclude the possibility of significant fibrosis in a large proportion of patients. However, their positive predictive values are weaker, even when these tests are combined. Above all, they do not allow us to follow the evolution of the fibrosis stage over time. This is why liver biopsies remain indispensable for determining the stage and severity of hepatic fibrosis and monitoring its evolution. It is therefore essential to develop more precise, non-invasive methods for accurately assessing the extent of liver fibrosis. This is the objective of the FreSH national cohort, which uses conventional biological techniques and in which our patients will also be included.

The hypothesis behind this initial pilot study is that 68Ga-FAPI-46 PET/CT imaging, which targets fibroblast activating protein (FAP), could provide a precise assessment of the severity and stages of liver fibrosis, as well as its distribution throughout the liver volume, and could ultimately be a useful tool for non-invasive monitoring of patients undergoing treatment. This technique has already been validated for the detection of numerous cancers, including hepatocarcinomas, and is capable of assessing renal fibrosis (pilot study with 15 patients), with a good correlation to biopsy and a direct link to glomerular filtration rate.

Targeted receptor (FAP) data also strongly support our hypothesis:

* FAP expression is negligible in healthy livers and proportional to the degree of fibrosis in pathological livers.
* Low plasma FAP concentrations rule out the hypothesis of hepatic fibrosis. PAF inhibitors also represent a very promising avenue of therapeutic research in NASH.

The HEFITEP study will assess for the first time the discriminative power of 68Ga-FAPI-46 PET/CT for grading liver fibrosis with reference to centrally analyzed liver biopsy in patients biopsied for suspected or proven non-alcoholic steatohepatitis (NASH).

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with recent liver biopsy for suspected or confirmed NASH
2. Individuals of legal age, who have received full information on the organization of the research and have signed an informed consent form.
3. Person, affiliated to a social security scheme or beneficiary of such a scheme.
4. Person who has undergone a preliminary clinical examination appropriate to the research.
5. Histological stage of fibrosis obtained at biopsy in accordance with the planned numbers (an equivalent number of patients with histological stages >2 and ≤ 2 must be recruited in each center, and a number of at least 16 patients must be included by all centers in each of the 4 groups of histological stages of fibrosis).

Exclusion Criteria:

1. Known hypersensitivity to 68Ga-FAPI-46 or to any of the excipients or components of the radiopharmaceutical.
2. Infection with HCV/HBV.
3. Decompensated cirrhosis (ascites, hepatic insufficiency, hepatorenal syndrome, etc.).
4. Known hepatocellular carcinoma.
5. Steatogenic treatment (corticosteroid, Tamoxifen, Amiodarone, Methotrexate).
6. Excessive alcohol consumption in the last 5 years (>210 g/week in men, >140 g/week in women).
7. Clinically unstable state not suitable for 68Ga-FAPI-46 PET/CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Capture intensity measurement | 1 year
  Measurement of 68Ga-FAPI-46 uptake intensity, with standardized uptake values in areas centred on the biopsy sites, the reference then being a classification of fibrosis stages determined by centralized biopsy rereading

SECONDARY OUTCOMES:
Standardized Uptake Value threshold values associated with each of the four fibrosis histological stage groups | 1 year
  Standardized Uptake Value threshold values associated with each of the four fibrosis histological stage groups (stages 4, 3, 2 and < 2) by the naive Bayes classifier.
Localization of the capture zone with maximum activity | 1 year
  Localization of the capture zone with maximum activity (SUVmax and SUV pic zones, respectively)
Search, on whole-body images, for 68Ga-FAPI-46 uptake | 1 year
  Search, on whole-body images, for 68Ga-FAPI-46 uptake foci located outside the tracer's normal elimination zones (urinary excretory tracts), and which may correspond to abnormal areas of fibrosis and/or inflammation, or even cancer
Intra-class correlation coefficients | 1 year
  Intra-class correlation coefficients and their 95% confidence intervals.
Variation in the degree of prediction of the four groups of histological stages of fibrosis | 1 year
  Variation in the degree of prediction of the four groups of histological stages of fibrosis when variables from 68Ga-FAPI-46 PET/CT are added to variables from usual clinical-biological scores